CLINICAL TRIAL: NCT06191835
Title: Implementation of a New Model of Care for Supporting Adherence in People Starting a New Medication for a Long-term Condition (myCare Start-I Project) - An Implementation Science Study - Phase A
Brief Title: Implementation of a New Model of Care for Supporting Long-term Medication Adherence (Phase A)
Acronym: myCareStart-I
Status: Active, not recruiting | Type: Observational
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: University of Basel (Other); Fundació Sant Joan de Déu (Other); pharmaSuisse, Switzerland (Unknown); Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other); University of Bern (Other)
Responsible Party: Principal Investigator, Marie Paule Schneider, PhD, Prof. Dr. Marie Paule Schneider, University of Geneva, Switzerland
Other Study IDs: 2023-01161
Record Dates: First submitted 2023-10-13; First posted 2024-01-05 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Medication Initiation for Long-term Conditions
Keywords: medication adherence; medication initiation; long-term treatment; implementation science; interprofessional collaboration; outpatient care; community pharmacy; General practitioner; cost-effectiveness; medication adherence support programme
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: myCare Start — The service consists of 2 times 10-minutes semi-structured pharmaceutical interventions between community pharmacist and patient, tailored to the patient's needs, positioned as partner, during the first 6 weeks after treatment initiation.
  Other Names: New Medicine Service

SUMMARY:
The overall objective of the myCare Start-I project is to adapt, implement and evaluate the myCare Start service within the Swiss pharmacy-physician network to enhance medication adherence during the initiation of a new long-term treatment. The study will use an implementation science approach. The myCare Start service is based on the New Medicine Service (NMS) that was developed in the United Kingdom.

DETAILED DESCRIPTION:
Phase A:

1. To conduct a contextual analysis of the current Swiss primary care ecosystem as related to pharmacy-physician interprofessional health services for patients with long-term diseases (i.e., contextual analysis).
2. To engage key stakeholders within the Swiss primary care ecosystem to contribute to the co-creation of a Swiss interprofessional myCare Start service (i.e., stakeholder involvement).
3. To design a contextually adapted myCare Start for use within Swiss community practice using contextually appropriate implementation strategies (i.e., intervention development/selecting implementation strategies).
4. To conduct feasibility testing on the contextually adapted intervention and implementation strategies and to develop an implementation research logic model (i.e., feasibility testing).

   Phase B: Please note Phase B will be carried out at a later date with further ethics committee approval.
5. To implement a contextually adapted Swiss myCare Start intervention in the pharmacy-physician network community and evaluate it in terms of medication adherence and cost-effectiveness outcomes.
6. To evaluate implementation outcomes and the implementation pathway of myCare Start.

ELIGIBILITY:
Phase A: contextual analysis

Inclusion Criteria:

* Community pharmacists and technicians of 5 participating pharmacies in the French-speaking part of Switzerland and 5 in the German-speaking part of Switzerland
* Primary care physicians working in collaboration or in the neighbourhood of the participating pharmacies
* Patients with long-term treatments, who are a regular patients of the included pharmacies
* International research groups who have implemented NMS within their countries or similar interventions.

Exclusion Criteria:

* Patients not willing to participate
* Patients that do not speak French or German

Phase B: hybrid type 2 effectiveness-implementation study

Patients are eligible for the myCare Start-I phase B study if :

* They are taking part in the myCare Start service
* They have been newly prescribed one or more new long-term medications in accordance with one of the five defined long-term conditions (cardiovascular disease (incl. hypertension and thromboprophylaxis), diabetes, hyperlipidaemia, depression and respiratory illness (asthma, COPD))
* They are 18 years or older
* They have mandatory basic health insurance in Switzerland
* They are able to self-manage treatment (i.e. they live at home without any support to manage their medication, exception: patient uses a pill dispenser and fills it in by him-/herself).
* They understand language spoken by pharmacy staff and are able to read and understand study documents (ge, fr)
* They are able to understand and willing to consent to the myCare Start study (including the agreement on self-reported questionnaires and collection of health care data via their health insurance company)

Exclusion criteria:

• Patients participating or having participated in an education program about their disease or treatment in the last 3 months, led by healthcare providers such as physicians, nurses, pharmacists or other (e.g. education provided by nurses for type I diabetes patients).

myCare Start definition of a new medication:

A new medication is a medication that has not been previously dispensed to the patient. This includes one or more new medications for a new diagnosis and or new medications for pre-existing diagnosis of a long-term condition.

Operational definition of a new medication:

* Active ingredient is indicated for one of the five long-term conditions (cardiovascular disease (incl. hypertension and thromboprophylaxis), diabetes, hyperlipidaemia, depression and respiratory illness (asthma, COPD)).
* Patient has never had this active ingredient dispensed before or restarts an active ingredient after a period of interruption of at least 12 months.

The new active ingredient can be part of a combo preparation (e.g. a diuretic added to an ACE inhibitor into the same preparation)

* Patient has had no change in active ingredient but has an important change in treatment administration, such as:

  * Change of galenic form (e.g. two different types on inhalators for asthma/COPD)
  * Intensification of dosage regimen (e.g. twice a day instead of once a day)
* The following change is not considered as medication initiation:

  * New dosage of already known active ingredient (e.g. dose escalation of antidepressants)
  * Simplification of administration mode (e.g. metformin 1000mg 1-0-0 instead of 500mg 1-0-1; change in antihypertensive drug regimen in elderly patients having vertigo in the morning: 0-0-X instead of X-0-0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phase A: contextual analysis
  Community pharmacists and technicians General practitioners or internal medicine physicians Patients with a long-term treatment International research groups
  Phase B: effectiveness-implementation study Patients with a long-term treatment for five long-term conditions (cardiovascular disease (incl. hypertension and thromboprophylaxis), diabetes, hyperlipidaemia, depression and respiratory illness (asthma, COPD))
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Medication adherence (objective measure) | 6 - 12 months
  Prescription renewal records (objective measure):
  Medication renewal records will be extracted from pharmaceutical records and analyzed using the "AdhereR" software in R.
Medication adherence (subjective measure) | 6 - 12 months
  Patient self-assessment (subjective measure):
  We will use the BAASIS© (Basel Assessment of Adherence to Immunosuppressive Medications Scale), a 6-item scale with demonstrated psychometric properties in transplantation and other chronic diseases, as it assesses adherence according to the ABC taxonomy (Initiation, Medication Implementation, and Persistence.
  The BAASIS scale has a minimum and maximum value of 6 and 30, respectively. Lower scores on the BAASIS indicate poorer adherence to immunosuppressive medications, while higher scores indicate better adherence. This self-report instrument consists of six items that assess different aspects of medication adherence, including dose taking, drug holidays, timing deviation, reduction of dose, persistence, and timing of dose taking.
Cost-effectiveness short-term | 12 months
  Total healthcare utilisation, in terms of total costs per patient, will be evaluated over the duration of the myCare Start follow-up period (12 months) using health insurance data. This will be combined with adherence results to determine the incremental cost-effectiveness ratio between the total costs per patient in the intervention vs. the control groups and the difference in adherence between groups. The survey will be forwarded to the patient at 14 days, 6 months, and 12 months after inclusion into the study via an emailed online survey.
  The main analysis consists of calculating 1) the incremental cost-effectiveness ratio between the total costs per patient in the intervention vs. the control group and 2.) the difference in adherence between groups and the probability that the intervention is cost-effective when the willingness to pay varies (i.e. the cost-effectiveness acceptability curve), the two classic indicators of cost-effectiveness analyses of health programmes.
Cost-effectiveness long-term | 12 months
  Long-term potential healthcare cost savings will be evaluated using Markov Modelling. The Markov Modelling approach applied in this study is an adapted version of the models previously used in the UK to evaluate the New Medicine Service, adjusted with parameters tailored to the Swiss context. This approach will enable the projection and estimation of medium- and long-term benefits arising from improved adherence to the prescriptions as a result of the myCare start intervention. In Switzerland, the most commonly prescribed medications for long-term illnesses include cholesterol-lowering therapies, type 2 diabetes drugs, hypertension treatments, and antidepressants. For these four medication groups, specific Markov models have been developed. These calculations will be conducted during the 12-month longitudinal follow-up phase.
Implementations Outcomes | 12 months
  The myCare start service will be evaluated in terms of acceptability, adoption, appropriateness, fidelity, feasibility, and implementation cost as proposed by Proctor's Implementation Outcomes Taxonomy (Proctor et al., 2019).
  Cost of implementation will be assessed using the time-driven activity-based cost (TDABC) instrument. This pragmatic method allows investigators to systematically estimate the cost of implementation strategies (e.g. training, reorganisation of practice, regular stakeholder meetings) and the cost of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Paule Schneider, PhD, Principal Investigator — University of Geneva
Locations (2):
- Switzerland (2):
  - Université de Genève, Geneva, Canton of Geneva
  - University of Basel, Basel

IPD SHARING:
Plan to Share IPD: Undecided
Once fully anonymized, quantitative data will be annotated and structured to make them sharable, and registered in a FAIR-compliant data repository.